CLINICAL TRIAL: NCT01465932
Title: Evaluation of the Effectiveness of Physical Therapy Program to Treat Rotator Cuff Disorders Among Nursing Professionals According to Indicators of Quality of Life and Job Satisfaction
Brief Title: Effectiveness of Physical Therapy Program to Treat Rotator Cuff Disorders Among Nursing Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Lisandra Vanessa Martins, Lisandra Vanessa Martins, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: uspombro01
Record Dates: First submitted 2011-10-25; First posted 2011-11-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-10

CONDITIONS: Shoulder Impingement Syndrome; Quality of Life; Satisfaction
Keywords: Nursing staff; Physical Therapy (Specialty)
MeSH Terms: conditions — Shoulder Impingement Syndrome; Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No proprioception (Active Comparator): Nursing professionals to diagnose disorders of the rotator cuff previously randomly allocated in this group did stretching exercises of the muscles of the cervical spine and chest, strengthening the muscles of the rotator cuff and stabilizers of the scapula, in addition to cryotherapy reduction of pain.
  Interventions: Other: Control, no Proprioception
- Proprioceptive exercises (Experimental): Nursing professionals to diagnose disorders of the rotator cuff previously randomly allocated in this group did stretching exercises of the muscles of the cervical spine and chest, strengthening the muscles of the rotator cuff and stabilizers of the scapula, proprioception exercises to improve motor control, besides cryotherapy for reduction of pain.
  Interventions: Other: Experimental, Proprioceptive exercises

INTERVENTIONS:
Other: Control, no Proprioception — The period of data collection period was from June 2010 to August 2011. All subjects who met the inclusion criteria, were randomly allocated to group 1 (control) or group 2 (experimental). Both groups consisted of 12 physical therapy sessions, taking place 2 times a week for 6 weeks. After randomization, subjects were allocated to group 1 (control group) underwent cervical stretching exercises, strengthening the scapular muscles and rotator cuff and cryotherapy.
  Other Names: No proprioception
  Arms: No proprioception
Other: Experimental, Proprioceptive exercises — The period of data collection period was from June 2010 to August 2011. All subjects who met the inclusion criteria, were randomly allocated to group 1 (control) or group 2 (experimental). Both groups consisted of 12 physical therapy sessions, taking place 2 times a week for 6 weeks. After randomization, subjects were allocated to group 2 (experimental group) underwent cervical stretching exercises, strengthening the scapular muscles and rotator cuff exercises and cryotherapy as well as proprioceptive sensory-motor
  Other Names: Proprioceptive exercises
  Arms: Proprioceptive exercises

SUMMARY:
The program of stretching, strengthening and proprioception is more effective than stretching and strengthening program in nursing, with rotator cuff disorder, according to indicators of quality of life and job satisfaction.

DETAILED DESCRIPTION:
The study will be conducted at the Rehabilitation Centre of the Hospital of the Medical School of Ribeirão Preto, University of São Paulo (USP-HCFMRP).

The study will be conducted with nursing staff (nurses, technicians and nursing assistants) HCFMRP-USP.

The sample will consist of nursing workers sent by request for referral to a medical diagnosis of rotator cuff disorder in the period May 2010 to August 2011.

There was no sample size calculation for this study because the number of subjects directly depends on the demand of patients referred to the Department of Physical Therapy Rehabilitation Center (CER) in the period of data collection. All patients who met the study inclusion criteria were invited to participate.

So, once met the inclusion criteria of the sample, the subjects were randomly allocated to Group 1 (control) or 2 (experimental).

Group 1 was formed by the subjects in the control group in which they were performed stretching exercises, cryotherapy and strengthening the shoulder.

Group 2 was formed by the subjects in the experimental group were performed in which stretching exercises, strengthening, and cryotherapy proprioceção shoulder.

ELIGIBILITY:
Inclusion Criteria:

* working as a nurse
* technician or nursing assistant in the hospital
* make medical diagnosis of disorder in the rotator cuff (impingement, injury or rupture of the cuff)
* does not make a medical diagnosis of cognitive impairment
* were receiving no another type of treatment for shoulder pain (eg medicines,acupuncture, massage)
* availability and interest in participating in therapy and accept to participate in the survey.

Exclusion Criteria:

* patients with pain that would prohibit their participation in the program with a medical diagnosis of cognitive impairment,
* associated with debilitating diseases,
* previous surgery of the shoulder,
* other specific conditions of the shoulder joint (adhesive capsulitis,
* degenerative osteoarthritis of the glenohumeral joint,
* tendon calcification) and do not accept to join the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Indicators of quality of life (WORC - Western Ontario Rotator Cuff The Index) | This scale is applied one day before and one day after the application of physical therapy intervention programs
  The WORC was selected to be a reliable tool for measuring quality of life for patients with rotator cuff disorder,available in Portuguese and validated for Brazilian culture by Lopes et al (2008).
  The WORC consists of 21 items and has five fields, and you can get the total for each domain separately. The domains are: physical symptoms, sports and recreation, work, lifestyle and emotions. The total score ranges from zero to 2100. Thus, zero implies no reduction in quality of life and the worst score is 2100.

SECONDARY OUTCOMES:
Questionnaire used was the Job Satisfaction Scale - Occupational Stress Indicator (OSI). | This scale is applied one day before and one day after the application of physical therapy intervention programs
  This scale allows for the measurement of satisfaction with 22 aspects of psychosocial work using Likert scales of six points, ranging from huge to enormous satisfaction dissatisfaction. Such a tool available in Portuguese was validated by Cooper, Sloan and Williams (1988).
  The sum of these measures provides an indicator of job satisfaction given by a global score that ranges from 22 to 123 points. There's a cutoff point defined herein

CONTACTS AND LOCATIONS:
Overall Officials: Lisandra V. Martins, postgraduate, Principal Investigator — University of Sao Paulo; Maria HP Marziale, Study Director — University of Sao Paulo
Locations (1):
- Hospital of Clinics, University of Medicine of Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Martins LV, Marziale MH. Assessment of proprioceptive exercises in the treatment of rotator cuff disorders in nursing professionals: a randomized controlled clinical trial. Rev Bras Fisioter. 2012 Nov-Dec;16(6):502-9. doi: 10.1590/s1413-35552012005000057. Epub 2012 Nov 2. PMID 23117648